CLINICAL TRIAL: NCT00960895
Title: Observational Study of Patients With Lymphangioleiomyomatosis and Pulmonary Hypertension
Brief Title: Pulmonary Hypertension in Lymphangioleiomyomatosis
Acronym: LAM-PH
Status: Completed | Type: Observational
Sponsor: Groupe d'Etudes et de Recherche sur les Maladies Orphelines Pulmonaires (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Vincent COTTIN, Pr Cottin, Groupe d'Etudes et de Recherche sur les Maladies Orphelines Pulmonaires, Groupe d'Etudes et de Recherche sur les Maladies Orphelines Pulmonaires
Other Study IDs: GERMOP-001
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Lymphangioleiomyomatosis; Pulmonary Hypertension
Keywords: Lymphangioleiomyomatosis; Pulmonary hypertension
MeSH Terms: conditions — Lymphangioleiomyomatosis; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a descriptive study of patients with Lymphangioleiomyomatosis and precapillary pulmonary hypertension.

DETAILED DESCRIPTION:
Descriptive study of patients with Lymphangioleiomyomatosis and precapillary pulmonary hypertension This will include modality of diagnosis of lLymphangioleiomyomatosis, results of right-sided heart catheterization, and pulmonary function tests

ELIGIBILITY:
Inclusion Criteria:

* Lymphangioleiomyomatosis (definite or probable), either sporadic or associated with tuberous sclerosis
* Precapillary pulmonary hypertension, as defined by right-sided heart catheterization (mean pulmonary artery pressure higher than 25 mmHg, wedge capillary pulmonary pressure less than 15 mmHg, pulmonary vascular resistance higher than 3 Wood units)

Exclusion Criteria:

* Post capillary pulmonary hypertension
* Other identifiable causes of pulmonary hypertension (ex: thromboembolic disease)
* Not willing to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lymphangioleiomyomatosis, either sporadic or associated with tuberous sclerosis Precapillary pulmonary hypertension, as defined by right-sided heart catheterization (mean pulmonary artery pressure higher than 25 mmHg, wedge capillary pulmonary pressure less than 15 mmHg, pulmonary vascular resistance higher than 3 Wood units)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Cottin, MD, Principal Investigator — University of Lyon
Locations (1):
- Louis Pradel Hospital, Lyon, University of Lyon, France